CLINICAL TRIAL: NCT01281020
Title: A 3-month, Observational Study Investigating With Electronic Monitoring the Level of Adherence and Treatment Satisfaction With Latanoprost/Timolol Fixed Combination Versus Unfixed Therapy in Open-angle Glaucoma
Brief Title: Adherence With Fixed Versus Unfixed Glaucoma Therapy
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Other Study IDs: NIS50/01/08
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Primary Open-angle Glaucoma; Ocular Hypertension; Exfoliation Glaucoma
Keywords: Glaucoma; Adherence; Fixed combination therapy
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Exfoliation Syndrome; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment with fixed combination: Patients who receive treatment with latanoprost/timolol fixed combination
- Treatment with unfixed therapy: Patients who receive latanoprost and timolol therapy

SUMMARY:
A 6-month, parallel, non-interventional trial investigating the level of adherence and the impact of dosing in open-angle glaucoma patients who receive either unfixed therapy with latanoprost once in the evening and timolol twice daily, or latanoprost/timolol fixed combination therapy once in the evening. All patients participating in this observational study will be monitored for their adherence with the use of Medication Event Monitoring System (MEMS). At the end of treatment periods treatment satisfaction will be assessed with selected questions from the Treatment Satisfaction Survey-Intraocular Pressure survey. This study will monitor objectively, for the first time, adherence and intraocular pressure control with fixed versus unfixed therapy. Finally it will help us to elucidate the impact of dosing (once-a-day versus three-times-daily) on the level of adherence in glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 21-80 years old
* Patient has ocular hypertension or open-angle glaucoma Patient receives therapy and is well controlled on fixed or unfixed latanoprost and timolol therapy
* Untreated IOP >19 mm Hg <33 mm Hg at baseline (10:00 hour)
* Open normal appearing angles
* Patient had at least a 20% reduction vs untreated baseline on current therapy
* Patient has early or moderate glaucoma (< 14 decibel; 0.8 or better cupping)
* Distance best corrected Snellen visual acuity greater than 1/10

Exclusion Criteria:

* Contraindication to timolol or prostaglandin therapy
* History of lack of response to any medication (< 10%)
* Patient does not understand the instructions and will not comply to medications
* Patient can not attend follow up
* Patient is a female of childbearing potential, or lactating mother
* History of trauma, inflammation, surgery, past use of steroids (within 2 months), severe dry eyes and use of contact lenses
* Sign of ocular infection
* A corneal abnormality that may affect IOP measurements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who use latanoprost/timolol fixed combination therapy with once-a-day dosing in the evening
  All patients already treated with timolol twice daily and latanoprost once in the evening
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Rate of adherence | 6 months
  Rate of asherence with fixed vs unfixed glaucoma therapy

SECONDARY OUTCOMES:
Ocular surface evaluation | 6 months
  Objective and subjective signs of ocular surface health
Treatment satisfaction | 6 months
  To document satisfaction with therapy this study will employ questions selected from a validated treatment satisfaction questionnaire (questions 10-15, Treatment Satisfaction Survey-Intraocular Pressure) as published by Day et al (Eye 2006; 20: 583-590). The survey will assess the level of satisfaction and overall quality-of-life with latanoprost/timolol fixed combination versus unfixed therapy in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios G Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, 1st University Department of Ophthalmology
Locations (1):
- Glaucoma Unit, 1st University Department of Ophthalmology, AHEPA Hospital, Thessaloniki, Greece